CLINICAL TRIAL: NCT05016999
Title: Evaluation of the Effect of the Consumption of a Combination of Allium Extracts on the Intestinal Microbiota in Healthy Elderly Resident Volunteers. Preliminary Study.
Brief Title: Allium Extracts on the Intestinal Microbiota in Healthy Resident Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DOMCA S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: C004
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2021-08

CONDITIONS: Intestinal Bacteria Flora Disturbance
Keywords: Garlic; Onion; Microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each volunteer is assigned a "participant number" that is associated with the "pot number" that contains the product that the volunteer must take.
  The "pot number" is the same as the "participant number". The pot does not indicate what product it is carrying.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Volunteers in this group will not take any products.
- Intervention (Experimental): Garlic concentrated extract plus onion concentrated extract plus microcrystalline cellulose (9892- Capsules®) up to 400 mg.
  Interventions: Dietary Supplement: Garlic and onion concentrate

INTERVENTIONS:
Dietary Supplement: Garlic and onion concentrate — Garlic extract concentrate (equivalent to 2 garlic cloves) and onion extract concentrate (equivalent to 1 onion)
  Other Names: AlioCare
  Arms: Intervention

SUMMARY:
To evaluate the effect of daily consumption of a combination of garlic and onion extracts on the intestinal microbiota and the production of short chain fatty acids in elderly healthy volunteers living in a residence.

Likewise, any incident related to health that occurred during that period will be noted.

DETAILED DESCRIPTION:
This study is a continuation of another (C002, registration number NCT04647071).

The volunteers from study C002 were invited to participate in this new study and, by the end of C002, all gave 2 stool samples.

After 4 weeks of washout, the control group volunteers in C002 will begin consuming 1 capsule per day of garlic and onion extract after lunch. The intervention group volunteers in C002 will not consume anything.

During 36 weeks any incident related to the health of the volunteers will be noted. Likewise, during this time, the volunteers will maintain their lifestyle and eating habits.

At 36 weeks, 2 stool samples will be taken from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years or older who participated in study C002.
* 2. Living in the Claret Residence for the Elderly in Granada during the study.
* Accept being vaccinated for the flu.
* Freely accepted to participate in the study and sign the informed consent document.
* Have the consent of the family.

Exclusion Criteria:

* Having any disease that affects the development and results of the study.
* Be unable to understand the study and sign voluntarily and freely the informed consent.
* Have a low expectation of compliance with the study protocol.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in bacterial species in feces. | 36 weeks.
  The bacterial populations present in the stool samples taken at the beginning and at the end of the study will be studied.
Short chain fatty acids in stool. | 36 weeks.
  Short chain fatty acids present in stool samples taken at the beginning and end of the study will be studied.

SECONDARY OUTCOMES:
Events during 36 weeks. | 36 weeks
  Any health-related events that occurred during the study and their duration will be noted.
Medication during 36 weeks. | 36 weeks
  The consumption of drugs during the study and its duration will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gracián Alcaide, MD, Principal Investigator — Claret Residence for the Elderly (Granada, Spain).
Locations (1):
- Residencia de Mayores Claret, Granada, Spain